CLINICAL TRIAL: NCT04402320
Title: Comparative Study Between Usage of NIV Versus MV for One Hour After Fulfillment of Weaning Criteria From Ventilation on Re-intubation in Post-traumatic ARDS
Brief Title: Non Invasive and Invasive Ventilation Post Extubation
Status: Completed | Type: Observational
Sponsor: King Abdul Aziz Specialist Hospital (Network)
Responsible Party: Sponsor
Other Study IDs: ICU-19-20
Record Dates: First submitted 2020-05-20; First posted 2020-05-26 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Respiratory Failure With Hypoxia
Keywords: non invasive ventilation invasive ventilation ARDS
MeSH Terms: interventions — Midazolam; Ventilators, Mechanical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Control group: extubated and weaning from the ventilator and followed our routine protocol of management post extubation without mechanical ventilation or BIPAP machine
  Interventions: Drug: Midazolam; Device: ventilator
- Invasive ventilation group: reconnected to mechanical ventilator before extubation for one hour with sedation with midazolam 3-5 milligram/hour intravenous infusion to achieve score 0 or -1on Richmond Agitation - Sedation Scale (RASS). 20 minutes before the end of this hour midazolam infusion discontinued and patients awaked. Patient put on mechanical ventilation (MV) with the following parameters, FIO2 40%, pressure SIMV mode, PEEP 8 cmH2O, Pressure support 15 cmH2O, Respiratory rate 14/min, Peak inspiratory pressure (PIP) of 35 cmH2O. Then patients extubated and followed our previous protocol without the use of NIV.
  Interventions: Drug: Midazolam; Device: ventilator
- non invasive ventilation group: following the same previous protocol done after extubation with immediate connection to NIV with BIPAP mode for 1 hour and repeated every 12hours for 48 hours, BIPAP adjusted in our study by FIO2 40%, PEEP 8 cmH2O, Pressure support of 15 cmH2O.
  Interventions: Drug: Midazolam; Device: ventilator

INTERVENTIONS:
Drug: Midazolam — reconnected to mechanical ventilation before extubation for one hour with sedation with midazolam 3-5 milligram/hour intravenous infusion to achieve score 0 or -1on Richmond Agitation - Sedation Scale (RASS). 20 minutes before the end of this hour midazolam infusion discontinued and patients awaked. Patient put on mechanical ventilation (MV) with the following parameters, FIO2 40%, pressure SIMV mode, PEEP 8 cmH2O, Pressure support 15 cmH2O, Respiratory rate 14/min, Peak inspiratory pressure (PIP) of 35 cmH2O. Then patients extubated and followed our previous protocol without the use
  Other Names: dormicum
Device: ventilator — reconnected to mechanical ventilation before extubation for one hour with sedation

SUMMARY:
Patients and methods: It is a prospective double blind study done on total 300 patients. Admitted with respiratory failure ARDS due to severe lung contusion. All of them selected to be ventilated for one week or more. Patients were randomly allocated in one of three groups each group contain 100 patients. Group A considered control extubated and follow our routine protocol, patients of group B reconnected to mechanical ventilation before extubation for one hour. patients of Group C extubated and immediately connected to NIV with BIPAP mode for 1 hour every 12 hours for 24 hours. Results: There was significant reduction in the number of patients had deterioration in conscious level in all the duration of the study in patients of both groups B and C compared to group A. Also significant reduction in the number of patients had deterioration in clinical parameters of respiration in all the duration of the study in patients of both groups B and C compared to group A as regards high respiratory rate, desaturation and development of hyperdynamic circulation (tachycardia and hypertension). significant reduction in the number of patients had multiple quadrant parenchymatous infiltration in all the duration of the study in patients of both groups B and C compared to group A. significant reduction in the number of patients had marked limitation to FEV1, FVC and MVV in all the duration of the study in patients of both groups B and C compared to group A. Conclusion: Use of either NIV every 12 hours for 24 hours or MV for one hour after fulfillment of weaning criteria reduces reintubation and post-extubation respiratory failure and decrease the ICU stay in critically ill patients with resolving ARDS due to severe lung trauma.

DETAILED DESCRIPTION:
It is a prospective double-blind study done on total 300 patients. Admitted to King Abdulaziz specialist hospital in Taif, KSA. Between April 2019 and April 2020 with respiratory failure ARDS due to severe lung contusion with these criteria: hypoxic index less than 200, bilateral parenchymatous lung infiltrate, no any acute cardiac insult, failed to maintain SPO2 more than 90% with Non-Invasive Ventilation (NIV) or need of continuous NIV to maintain the previous saturation. This selected ARDS was due to lung contusion which diagnosed by Computerized tomography of the chest following chest trauma. All of them selected to be ventilated for one week or more and only those who showed full criteria of weaning from the ventilator enrolled in our study. Our criteria of weaning include fully conscious patients, hemodynamically stable without any inotropic support, hypoxic index(PAO2/FIO2) more than 200 calculated from the arterial blood gases (ABG), bicarbonate level in arterial blood more than 20 mmol/l, hemoglobin level more than 10 gm%, chest X ray less than one quadrant parenchymatous infiltration in each lung on Murray score of chest Xray, rapid shallow breathing index <105. Patients were randomly allocated in one of three groups each group contain 100 patients. Randomization sequence was created using Excel 2007 (Microsoft, Redmond, WA, USA) with a 1:1 allocation using random block sizes of 2 and 4 by an independent doctor. In this way, sequence generation and type of randomization can be expressed at the same time. Patients of group A extubated and followed our routine protocol of management post extubation which include Nebulization with Ventolin and epinephrine racemic every 8 hours for 48 hours, chest physical therapy (CPT) every 6 hours for 48 hours include clapping percussion with mechanical vibration and suction plus huffing or coughing and postural drainage if there was atelectasis seen by our routine chest X ray. Patients of group B reconnected to mechanical ventilation before extubation for one hour with sedation with midazolam 3-5 milligram/hour intravenous infusion to achieve score 0 or -1on Richmond Agitation - Sedation Scale (RASS). 20 minutes before the end of this hour midazolam infusion discontinued and patients awaked. Patient put on mechanical ventilation (MV) with the following parameters, FIO2 40%, pressure SIMV mode, PEEP 8 cmH2O, Pressure support 15 cmH2O, Respiratory rate 14/min, Peak inspiratory pressure (PIP) of 35 cmH2O. Then patients extubated and followed our previous protocol without the use of NIV.

ELIGIBILITY:
Inclusion Criteria:

* respiratory failure ARDS due to severe lung contusion

Exclusion Criteria:

* post arrest, deeply comatosed patients and children below 18 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — adult only 18-65 years
Study Population: on total 300 patients. Admitted to King Abdulaziz specialist hospital in Taif, KSA. Between April 2019 and April 2020 with respiratory failure ARDS due to severe lung contusion with these criteria: hypoxic index less than 200, bilateral parenchymatous lung infiltrate, no any acute cardiac insult, failed to maintain SPO2 more than 90% with Non-Invasive Ventilation (NIV) or need of continuous NIV to maintain the previous saturation. This selected ARDS was due to lung contusion which diagnosed by Computerized tomography of the chest following chest trauma. All of them selected to be ventilated for one week or more and only those who showed full criteria of weaning from the ventilator enrolled in our study
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
number of patients re-intubated within 48 hours and shorten the duration of ICU stay | 48 hours
  monitoring hemodynamics, oxygenation, and conscious level in the studied duration

CONTACTS AND LOCATIONS:
Locations (1):
- King abd el Aziz specialist hospital, Ta'if, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
see if both iv or niv after fullfilling the criteria of extubation in ARDS patients can prevent reintubation